CLINICAL TRIAL: NCT00458250
Title: Haploidentical Hematopoietic Stem Cell Transplantation in the Treatment of Hematological Malignancies Using CAMPATH-1H
Brief Title: Feasibility of Haploidentical Hematopoietic Stem Cell Transplantation Using CAMPATH-1H
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Tehran University of Medical Sciences (Other)
Allocation: Non-Randomized | Model: Factorial | Masking: None | Purpose: Treatment
Other Study IDs: 418-A-1954
Record Dates: First submitted 2007-04-07; First posted 2007-04-10 (Estimated); Last update posted 2008-11-18 (Estimated); Status verified 2008-11

CONDITIONS: Leukemia, Myeloid, Acute; Leukemia, Lymphoblastic, Acute
Keywords: Hematopoietic Stem Cell Transplantation; Haploidentical; Hematologic Neoplasms; human, Bone Marrow; Granulocyte Colony-stimulating Factor; CAMPATH; Alemtuzumab; AML; ALL; 10. Eligibility
MeSH Terms: conditions — Leukemia, Myeloid, Acute; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Hematologic Neoplasms | interventions — Busulfan; Cyclophosphamide; Alemtuzumab; Cyclosporine; Methotrexate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Procedure: Haploidentical hematopoietic stem cell transplantation
Drug: Busulfan
Drug: Cyclophosphamide
Drug: CAMPATH-1H
Drug: Cyclosporin A
Drug: Methotrexate

SUMMARY:
Many patients suffering various malignant and non-malignant diseases need hematopoietic stem cell transplantation from a healthy person. In the majority of cases there is no matched related or unrelated donor.

Some researchers have been performed transplantation from semi-matched (haploidentical) related donors with relatively good results.

Chinese researchers have been performed this kind of transplantation using CAMPATH-1H and their reports indicates good results.

Chinese populations have more homogenous genetic background than Iranians. In this project, we are going to study the feasibility of this method of haploidentical transplantation in Iranian patients.

DETAILED DESCRIPTION:
Haploidentical hematopoietic stem cell transplantation is a very important therapeutic intervention for treatment of some genetic disorders and hematological malignancies.

In the majority of cases, there is no matched related or unrelated donor. Haploidentical hematopoietic stem cell transplantation is a promising alternative for critical cases.

To avoid severe graft versus host disease (GVHD), two types of T cell depletion (TCD) had been used: total TCD and partial TCD.

Total TCD has disadvantages such as increased rate of rejection and relapse, and increased rate of infections due to delayed immune reconstitution.

Partial TCD has been done by in vivo and/or in vitro methods. In haploidentical transplantation, donor partial TCD (ex vivo TCD) without recipient TCD increases the rate of rejection and can not prevent severe GVHD successfully.

In vivo TCD by partial depletion of donor and recipient T cells has been done in haploidentical transplantation with good results (to some extent inferior to full matched transplantations) by using CAMPATH, ATG, etc.

Most of these studies have been performed in Chinese and Japanese populations that have more homogenous genetic background than other populations.

In order to study the feasibility of this kind of transplantation in Iranian patients, we defined a project to perform haploidentical hematopoietic stem cell transplantation by using in vivo CAMPATH-1H.

ELIGIBILITY:
Inclusion Criteria:

INCLUSION CRITERIA - RECIPIENT: (all of the following)

* Ages 5-50 years
* Acute myelogenous leukemia (AML) or acute lymphoblastic leukemia (ALL)
* Second remission (CR2) in standard risk patients or CR1 in cases with high-risk features (poor cytogenetic changes or secondary to myelodysplastic syndrome)
* Unavailability of HLA identical related donor or matched unrelated donor.
* Unavailability of other therapeutic intervention that prolongs patient survival.
* Lack of active infection.
* No history of allergy to CAMPATH.
* For adults: Ability to comprehend the investigational nature of the study and provide informed consent. For minors: Written informed consent from one parent or guardian..
* Social and intellectual competency of the patient and his/her family to follow medical recommendations.

INCLUSION CRITERIA - DONOR:

* The donor must be haploidentical with the recipient: In the order of priority, siblings who have an identical paternal HLA haplotype with the patient, offspring (for female patients that do not have appropriate sibling), and mother.
* Possibly, it is better that the donor and recipient to be of same blood group and sex..
* Possibly, it is better that female donors not to be multiparous.
* Weight greater than or equal to 18 kg.
* Age between 2 and 60 years old.
* For adults: Ability to comprehend the investigational nature of the study and provide informed consent. For minors: Written informed consent from one parent or guardian and informed assent: The process will be explained to the minor on a level of complexity appropriate for their age and ability to comprehend.
* Negative two-way WBC crossmatch with the recipient.

Exclusion Criteria:

EXCLUSION CRITERIA - RECIPIENT: (ANY OF THE FOLLOWING)

* Major anticipated illness or organ failure incompatible with survival from transplantation.
* Severe psychiatric illness. Mental deficiency sufficiently severe as to make compliance with the transplantation procedure unlikely and making informed consent impossible.
* Positive pregnancy test for women of childbearing age.
* HIV positive
* Active infection
* Left ventricular ejection fraction less than 40%
* AST/SGOT greater than 20 x ULN (CTCAE grade IV v3.0)
* Bilirubin greater than 10 x ULN (CTCAE grade IV v3.0)
* Creatinine greater than 6 x ULN (CTCAE grade IV v 3.0)
* Occurrence of allergy symptoms and signs during CAMPATH infusion. EXCLUSION CRITERIA - DONOR: (ANY OF THE FOLLOWING)
* Pregnant or lactating
* Unfit to receive filgrastim (G-CSF) and undergo apheresis (abnormal blood counts, history of stroke, uncontrolled hypertension)
* Sickling hemoglobinopathies including HbSS, HbAS, HbSC
* HBsAg or HIV positive
* Active infection
* CMV positive (for CMV negative recipients)
* Severe psychiatric illness. Mental deficiency sufficiently severe as to make compliance with the BMT treatment unlikely and making informed consent impossible
* Contraindication to general anesthesia.

Ages: 2 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 10 (Estimated)
Dates: Start 2006-09; Study Completion 2008-02 (Actual)

PRIMARY OUTCOMES:
Engraftment one month after transplantation | Up to 30 days from transplantation

SECONDARY OUTCOMES:
six months survival | Up to 180 days after transplantation

CONTACTS AND LOCATIONS:
Overall Officials: Mohammadreza Ostadali, MD, Ph.D., Study Director — Hematology-Oncology & BMT Research Center; Ardeshir Ghavamzadeh, MD, Principal Investigator — Hematology-Oncology & BMT Research Center; Kamran Alimoghaddam, MD, Principal Investigator — Hematology-Oncology & BMT Research Center
Locations (1):
- Hematology-Oncology & BMT Research Center, Tehran, Tehran Province, Iran